CLINICAL TRIAL: NCT01903850
Title: A PROSPECTIVE, MULTI-CENTER PILOT STUDY OF THE truFREEZE™ SYSTEM TO ASSESS THE EFFICACY AND SAFETY OF CRYO SPRAY ABLATION IN THE TREATMENT OF AIRWAY OBSTRUCTIONS (TruFreeze AIRWAY OBSTRUCTION - "TAO" STUDY)
Brief Title: TruFreeze™ Airway Obstruction: TAO STUDY
Acronym: TAO
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawn for business reasons
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CSA 005
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Lung Disease Airways; Lung Diseases, Obstructive; Airway; Obstruction, With Emphysema; Airway Obstruction
Keywords: Benign central airway obstruction; Malignant central airway obstruction; Spray cryotherapy; Endoluminal tumors; Airway granulation tissue
MeSH Terms: conditions — Lung Diseases, Obstructive; Bites and Stings; Airway Obstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- spray cryotherapy (Experimental): spray cryotherapy: 4 -5 second sprays at Baseline (possible additional tx. to be determined at follow up)
  Interventions: Device: spray cryotherapy

INTERVENTIONS:
Device: spray cryotherapy — spray cryotherapy
  Other Names: truFreeze™ Spray cryotherapy

SUMMARY:
The purpose of this study is to prospectively assess the efficacy and safety of spray cryotherapy ablation with the truFreeze System in conjunction with mechanical dilation or debridement for the treatment of clinically significant obstructions of the central airways. The primary effectiveness endpoint is the proportion of subjects with a minimum of 25% improvement in luminal patency following SCT treatment and mechanical intervention 30 days (+/- 5 days) following treatment. Additionally, a primary clinical safety endpoint is the reporting of all adverse events.

DETAILED DESCRIPTION:
This multi-center prospective feasibility study will enroll at up to 6 clinical sites for a total of 30 subjects. Enrollment criteria includes subjects with clinically significant benign or malignant obstructions of the central airways, who require treatment intervention and are not candidates for surgical resection. The central airways are defined as including the trachea, left or right main bronchus, or the bronchus intermedius on the right. Spray cryotherapy (SCT) using the truFreeze system will be used in conjunction with mechanical interventions (balloon/rigid dilation or debridement of tumors) to improve airway patency. Subjects will receive up to 4, 5-second spray cycles prior to mechanical intervention (balloon/rigid dilation or debridement of tumors), followed by up to 4, 5-second additional spray cycles immediately following mechanical intervention.

The degree of airway narrowing will be estimated by the treating physicians before and after each treatment using a graded scale. Digital endoscopic images of each obstruction taken before and after each treatment, will also be assessed by a neutral assessor blinded to treatment. Subjects will be contacted on Day 1 following treatment to assess for any treatment related adverse events. Subjects may undergo a repeat bronchoscopy two weeks (14 days +/- 2 days) following the initial SCT treatment if clinically indicated or routine practice of the treating physician. A SCT treatment at a NORMAL flow setting may be performed at the 14 day bronchoscopy if deemed clinically indicated. If subjects are treated with SCT at the 14-day treatment, they will again be contacted on Day 1 following treatment to assess for any treatment related adverse events.

A follow-up bronchoscopy to reassess luminal patency and treatment site healing response will be performed at 30 days (+/- 5 days) following the last SCT treatment. The last SCT treatment may be the initial treatment day or 14-day treatment if performed. again, the degree of airway narrowing will be estimated by the treating physicians using a graded scale and digital endoscopic images of each obstruction will be taken to be assessed by a neutral assessor blinded to treatment.

The primary efficacy endpoint for statistical analysis and study powering will be the proportion of subjects exhibiting an adequate (minimum of 25%) improvement in airway patency. Based on prior clinical experience with liquid nitrogen spray cryotherapy and other ablation techniques, a response rate of approximately 80% is anticipated. This study is powered to detect a 20% lower response rate (i.e. 60% or lower) compared to the expected rate.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with symptomatic, clinically significant central airway obstruction requiring treatment intervention and who are not candidates for surgical resection. The central airway obstruction must be a consequence of any of the following:

   1. Benign airway strictures
   2. Primary or secondary endobronchial tumors located in the central airways
   3. Airway stents complicated by significant granulation tissue
2. Subjects (or designated proxies) who are able to provide written informed consent
3. Subjects aged 18 years or greater
4. Subjects with Eastern Cooperative Oncology Group (ECOG) performance status of 3 or less
5. Subjects deemed eligible candidates for spray cryotherapy based on medical history and physical exam

Exclusion Criteria:

1. Subjects undergoing treatment with any other investigational therapy within the month preceding cryotherapy or planned within 1 month following treatment

   a. Subjects with malignant strictures who require chemotherapy/radiation therapy (including investigational therapies) within 30 days will be allowed participation in the study.
2. Subjects with extraluminal causes of airway obstruction such as bulky mediastinal adenopathy, or a central mediastinal tumor causing compression of the airway
3. Subjects with less than 3 month expected survival
4. Subjects who it is anticipated will require stent placement during their initial treatment
5. Subjects who are pregnant or nursing, per device instructions for use
6. Subjects (or a designated proxy) who are unwilling to provide written informed consent
7. Subjects with ECOG performance status greater than 3
8. Subjects likely to have difficulty complying with study visit follow-up scheduling
9. Known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up
10. Subjects with uncontrolled coagulopathy or other bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The primary clinical effectiveness endpoint is a minimum of 25% improvement in luminal patency following SCT treatment and mechanical intervention, on the Day 30 assessment following the last SCT treatment. | 30 - 44 Days (+/- 5 days)
  The primary efficacy endpoint for statistical analysis and study powering is the proportion of subjects exhibiting an adequate (minimum of 25%) improvement in airway patency on the Day 30 assessment following the last SCT treatment.

SECONDARY OUTCOMES:
Subject symptoms and functional status | 30-44 days (+/- 5 days)
  Secondary endpoint will consist of a measure of changes in subject symptoms and functional status prior to and 30 days (+/- 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Hiran C Fernando, MD, Principal Investigator — Boston Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ernst A, Feller-Kopman D, Becker HD, Mehta AC. Central airway obstruction. Am J Respir Crit Care Med. 2004 Jun 15;169(12):1278-97. doi: 10.1164/rccm.200210-1181SO. PMID 15187010
- [Background] Johnston CM, Schoenfeld LP, Mysore JV, Dubois A. Endoscopic spray cryotherapy: a new technique for mucosal ablation in the esophagus. Gastrointest Endosc. 1999 Jul;50(1):86-92. doi: 10.1016/s0016-5107(99)70352-4. PMID 10385730
- [Background] Greenwald BD, Dumot JA, Horwhat JD, Lightdale CJ, Abrams JA. Safety, tolerability, and efficacy of endoscopic low-pressure liquid nitrogen spray cryotherapy in the esophagus. Dis Esophagus. 2010 Jan;23(1):13-9. doi: 10.1111/j.1442-2050.2009.00991.x. Epub 2009 Jun 9. PMID 19515183
- [Background] Shaheen NJ, Greenwald BD, Peery AF, Dumot JA, Nishioka NS, Wolfsen HC, Burdick JS, Abrams JA, Wang KK, Mallat D, Johnston MH, Zfass AM, Smith JO, Barthel JS, Lightdale CJ. Safety and efficacy of endoscopic spray cryotherapy for Barrett's esophagus with high-grade dysplasia. Gastrointest Endosc. 2010 Apr;71(4):680-5. doi: 10.1016/j.gie.2010.01.018. PMID 20363409
- [Background] Greenwald BD, Dumot JA, Abrams JA, Lightdale CJ, David DS, Nishioka NS, Yachimski P, Johnston MH, Shaheen NJ, Zfass AM, Smith JO, Gill KR, Burdick JS, Mallat D, Wolfsen HC. Endoscopic spray cryotherapy for esophageal cancer: safety and efficacy. Gastrointest Endosc. 2010 Apr;71(4):686-93. doi: 10.1016/j.gie.2010.01.042. PMID 20363410
- [Background] Xue HB, Tan HH, Liu WZ, Chen XY, Feng N, Gao YJ, Song Y, Zhao YJ, Ge ZZ. A pilot study of endoscopic spray cryotherapy by pressurized carbon dioxide gas for Barrett's esophagus. Endoscopy. 2011 May;43(5):379-85. doi: 10.1055/s-0030-1256334. Epub 2011 Mar 24. PMID 21437849
- [Background] Halsey KD, Chang JW, Waldt A, Greenwald BD. Recurrent disease following endoscopic ablation of Barrett's high-grade dysplasia with spray cryotherapy. Endoscopy. 2011 Oct;43(10):844-8. doi: 10.1055/s-0030-1256649. Epub 2011 Aug 8. PMID 21826629
- [Background] Fernando HC, Dekeratry D, Downie G, Finley D, Sullivan V, Sarkar S, Rivas R Jr, Santos RS. Feasibility of spray cryotherapy and balloon dilation for non-malignant strictures of the airway. Eur J Cardiothorac Surg. 2011 Nov;40(5):1177-80. doi: 10.1016/j.ejcts.2011.02.062. Epub 2011 Apr 8. PMID 21482131
- [Background] Krimsky WS, Rodrigues MP, Malayaman N, Sarkar S. Spray cryotherapy for the treatment of glottic and subglottic stenosis. Laryngoscope. 2010 Mar;120(3):473-7. doi: 10.1002/lary.20794. PMID 20058314
- [Background] Krimsky WS, Broussard JN, Sarkar SA, Harley DP. Bronchoscopic spray cryotherapy: assessment of safety and depth of airway injury. J Thorac Cardiovasc Surg. 2010 Mar;139(3):781-2. doi: 10.1016/j.jtcvs.2009.03.051. Epub 2009 Aug 6. No abstract available. PMID 19664781
- [Background] Finley DJ, Dycoco J, Sarkar S, Krimsky WS, Sherwood JT, Dekeratry D, Downie G, Atwood J, Fernando HC, Rusch VW. Airway spray cryotherapy: initial outcomes from a multiinstitutional registry. Ann Thorac Surg. 2012 Jul;94(1):199-203; discussion 203-4. doi: 10.1016/j.athoracsur.2012.01.112. Epub 2012 Apr 18. PMID 22516831
- [Background] Au JT, Carson J, Monette S, Finley DJ. Spray cryotherapy is effective for bronchoscopic, endoscopic and open ablation of thoracic tissues. Interact Cardiovasc Thorac Surg. 2012 Oct;15(4):580-4. doi: 10.1093/icvts/ivs192. Epub 2012 Jul 18. PMID 22811511